CLINICAL TRIAL: NCT07125287
Title: "Confront the Fear" - Evaluation of a Novel Exposure-Based CBT for Youth With Blood and Injection Phobia and Concurrent Somatic Illness Requiring Injections
Brief Title: Exposure-Based CBT for Youth With Blood and Injection Phobia and Chronic Illness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Charlotte S Gentili, Lic Psychologist, PhD, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-08344-01; K 2025-5350 (Other: Stockholm Region)
Record Dates: First submitted 2025-06-27; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Blood Injury Phobia; Injection Fear
Keywords: Phobia exposure; CBT; Needle exposure practice kit for home use
MeSH Terms: conditions — Iatrophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Exposure based CBT
  Interventions: Behavioral: Exposure based CBT

INTERVENTIONS:
Behavioral: Exposure based CBT — This intervention is an exposure-based CBT program developed for children with blood-injection-injury (BII) phobia and a co-occurring somatic illness. The treatment includes a structured home training kit with medical materials (e.g., syringes, swabs) related to the child's fear, enabling frequent and realistic exposure exercises at home between sessions, guided by parents. This allows for higher treatment intensity and continuity. The intervention is tailored to children who require regular medical procedures and whose phobia interferes with essential care. Unlike previous studies, this model integrates both clinical sessions and structured home practice to increase adherence and reduce fear in medical settings.

SUMMARY:
More than half of all children fear needles, and hospitalized children often describe injections as the most frightening part of medical care. While mild needle fear can often be managed by healthcare staff using distraction and reassurance, these strategies are ineffective for children with blood-injection-injury phobia (BII phobia). Children with BII phobia and co-occurring chronic medical conditions often require repeated blood tests or injections, but their phobia may prevent essential treatment. In such cases, healthcare providers may be forced to use physical restraint, sedation, or general anesthesia-approaches that are distressing for the child and costly for the healthcare system.

Although exposure-based cognitive behavioral therapy (CBT) is an effective treatment for specific phobias in adults, there is very limited research on CBT for children with BII phobia, particularly those with serious medical conditions. At the Department of Behavioral Medicine at Karolinska University Hospital, we have developed an exposure-based CBT intervention tailored for children with BII phobia and co-occurring somatic illness. The program includes a home-based training kit with medical materials to support frequent and realistic exposure between clinic sessions. Clinical experience suggests the intervention improves fear responses and increases medical treatment adherence, but it has not yet been formally evaluated.

This study aims to evaluate the feasibility and effectiveness of this novel CBT intervention for children and adolescents with disabling BII phobia and chronic somatic conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-17 years;
2. Blood-Injection-Injury (BII) phobia;
3. Somatic disease or condition requiring regular injections and/or blood sampling;
4. Ability to read and write in Swedish.

Exclusion Criteria:

1. Significant cognitive or intellectual impairment;
2. Severe psychopathology (e.g., suicidality);
3. Acute trauma;
4. Ongoing or recently completed treatment for BII phobia.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavior Avoidance Test (BAT) | Baseline (prior to treatment session 1) and post-treatment (at treatment session 11)
  An observational assessment in which the patient is asked to approach a feared situation or stimulus as far as they can, based on a predefined hierarchy of difficulty or anxiety levels. The BAT is commonly used to assess the degree of avoidance and fear in relation to specific phobia-related stimuli, and to evaluate treatment progress and outcomes. In this study, the BAT will be used to measure behavioral avoidance.
Injection Phobia Scale (IPS) | Baseline (at treatment session 1), post-treatment (at treatment session 11), and follow-up at 1 month and 3 months post-treatment
  A child-adapted version of the Injection Phobia Scale (Öst, Hellström & Kåver, 1992). In this study, only the subscale measuring anxiety level is used. The original subscale has demonstrated high internal consistency, with a Cronbach's alpha of 0.86. The scale consists of 18 items, each rated on a five-point scale where the respondent indicates the amount of fear they would experience in different situations.

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale 25 items (RCADS-25) | Baseline (at treatment session 1), post-treatment (at treatment session 11), and follow-up at 1 month and 3 months post-treatment
  The Revised Child Anxiety and Depression Scale (RCADS) is a standardized self-report questionnaire designed to assess symptoms of anxiety and depression in children and adolescents. It includes multiple subscales that measure various anxiety disorders (such as generalized anxiety, social phobia, separation anxiety, panic disorder, and obsessive-compulsive disorder) as well as depression symptoms. The RCADS is widely used in clinical and research settings due to its strong psychometric properties, including good reliability and validity. Respondents rate the frequency of symptoms on a Likert-type scale, providing a comprehensive profile of internalizing symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Kemani, PhD, Principal Investigator — Karolinska Universitetssjukhuset, Region Stockholm

IPD SHARING:
Plan to Share IPD: No
Due to ethical approval conditions and applicable data protection laws, individual participant data (IPD) will not be shared with other researchers.